CLINICAL TRIAL: NCT01900873
Title: Effects of Inspiratory Muscle Training on Dyspnea Perception During Exercise in Patients With COPD
Acronym: IMTCOCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Queen's University, Kingston, Ontario (Other)
Responsible Party: Principal Investigator, Daniel Langer, Postdoctoral Research Fellow Research Foundation Flanders, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMED-1579-13
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: COPD; Severe Systemic Illness-induced Respiratory Muscle Wasting
Keywords: Inspiratory Muscle Training; COPD; Inspiratory Muscle Function; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory Muscle Strength Training (Experimental): High intensity inspiratory muscle training
  Interventions: Device: Inspiratory Muscle Strength Training
- Inspiratory Muscle Endurance Training (Sham Comparator): Sham inspiratory muscle training at low intensity
  Interventions: Device: Inspiratory Muscle Endurance Training

INTERVENTIONS:
Device: Inspiratory Muscle Strength Training — IMT will be performed using a variable flow resistive loading device (POWERbreathe®KH1, HaB International Ltd., Southam, UK). The device is able to store training parameters of up to 40 sessions. Most training sessions during this RCT will be performed by patients at their homes without supervision. The intervention group (strength IMT) will perform two daily sessions of 30 breaths. Measurements of Pi,max will be performed every week and training loads will be increased continuously to maintain at least 40-50% of the actual Pi,max values. Each week, one training session will be performed under supervision. Training load will be increased during this session.
  Other Names: Electronic Variable Flow Resistive Loading IMT Device; POWERbreathe®KH1, HaB International Ltd., Southam, UK
  Arms: Inspiratory Muscle Strength Training
Device: Inspiratory Muscle Endurance Training — IMT will be performed using a variable flow resistive loading device (POWERbreathe®KH1, HaB International Ltd., Southam, UK). The device is able to store training parameters of up to 40 sessions. Most training sessions during this RCT will be performed by patients at their homes without supervision. The sham group (endurance IMT) will perform three daily sessions of 30 breaths and will train at a constant inspiratory load of no more than 10% of their initial Pi,max. Each week, one training session will be performed under supervision.
  Other Names: Electronic Variable Flow Resistive Loading IMT Device; POWERbreathe®KH1, HaB International Ltd., Southam, UK
  Arms: Inspiratory Muscle Endurance Training

SUMMARY:
Patients with chronic obstructive pulmonary disease are often limited in their exercise capacity by intolerable shortness of breath (dyspnea). Patients are breathing at high lung volumes during exercise which forces inspiratory muscles to work at a high percentage of their maximal capacity. This increased inspiratory effort has been shown to be independently related to symptoms of dyspnea during exercise in previous research. Eight weeks of high intensity variable flow resistive inspiratory muscle training is hypothesized to reduce inspiratory effort and to decrease neural drive to inspiratory muscles. These factors are hypothesized to jointly contribute to delaying the occurrence of intolerable symptoms of dyspnea and to improve exercise tolerance in these patients.

DETAILED DESCRIPTION:
We want to study whether a highly intense inspiratory muscle training program improves exercise capacity by reducing inspiratory effort, improving pulmonary mechanics and delaying the development of intolerable symptoms of dyspnea during cycle exercise. Eight weeks of high intensity variable flow resistive inspiratory muscle training is hypothesized to reduce inspiratory effort and to decrease neural drive to inspiratory muscles. The ratio of inspiratory effort to volume displacement should improve, and reductions of inspiratory capacity during exercise should be delayed. These factors are hypothesized to jointly contribute in delaying the occurrence of intolerable symptoms of dyspnea and to improve exercise tolerance in these patients.

We will study physiological mechanisms by which inspiratory muscle training exerts its effects on dyspnea reduction and exercise capacity. In this clinical trial patients will be randomly allocated into either an intervention or a control group. The intervention group will receive a highly intense inspiratory muscle training program that will improve inspiratory muscle function. The control group will receive a sham training that will not result in physiological benefits.

During the 8-week training period patients will have to attend the hospital once weekly for a short visit to perform a training session under supervision. Before the training intervention patients will be assessed twice and then again once after the 8-week program. This means that this trial will involve a total of 11 visits (3 long visits (approximately 4h) for assessments and 8 short visits (approximately 30 minutes) for supervised training sessions) over a period of 2-3 months. Assessments of pulmonary function, inspiratory muscle function, exercise capacity, daily physical activity and symptoms of dyspnea during exercise will be performed. Pulmonary mechanics and inspiratory muscle activation during exercise will also be assessed.

Stable COPD patients with pronounced inspiratory muscle weakness (Pi,max < 70cmH2O or <70% predicted) will be eligible to participate in the study. Exclusion criteria will be diagnosed psychiatric or cognitive disorders, progressive neurological or neuromuscular disorders and severe orthopedic problems having a major impact on exercise capacity.

Patients in both the intervention and the placebo group will follow an eight-week IMT program. They will receive either high intensity IMT (intervention group) or sham IMT (placebo group). Interventions will be presented to patients as strength training (intervention group) or endurance training (placebo group). Measurements of primary and secondary endpoints will be performed before and after 8 weeks of IMT. All tests will be performed by an experienced investigator that will be blinded to group allocation.

Total training load for both groups will be two to three daily sessions of 30 breaths (3-4 minutes per session), on 7 days per week, for 8 weeks. IMT will be performed using a variable flow resistive loading device(POWERbreathe®KH1, HaB International Ltd., Southam, UK).

Differences in primary and secondary outcomes between groups after 8 weeks of IMT will be compared adjusting for baseline differences in an analysis of covariance (ANCOVA).

Dyspnea perception on a 10-point Borg Scale (BORG CR10) at identical ventilation during the constant work rate cycling test after the intervention will be the primary outcome. To detect a difference of one point in the dyspnea perception on a 10-point Borg Scale at identical ventilation during the constant work rate cycling test after the intervention between subjects, assuming a standard deviation of the changes in dyspnea perception between baseline and follow-up measurement of 1 point with a degree of certainty (statistical power) of 80% and a risk for a type I error (a) < 5%, a sample size of 16 patients for each group is needed. These estimates are based on previous work on dyspnea perceptions during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of COPD
* Inspiratory Muscle Weakness (Pi,max < 70cmH2O or < 70% predicted)

Exclusion Criteria:

* Major cardiovascular, orthopedic, or cognitive impairments limiting exercise capacity more than pulmonary function impairment.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Dyspnea (Borg CR-10 scale) | Change from Baseline in Borg CR-10 scale at 8 weeks
  Numerical value reported for intensity of dyspnea (shortness of breath) ranging from 0 (no symptoms) to 10 (maximal symptoms)

SECONDARY OUTCOMES:
Maximal inspiratory pressure (Pi,max) | Change from Baseline in Pi,max at 8 weeks
  Maximal voluntary inspiratory pressure will be recorded at the mouth to assess inspiratory muscle strength (pressure generating capacity). Measurements will be performed at functional residual capacity for inspiratory respiratory pressure (maximal inspiratory pressure; Pi,max ) using the technique proposed by Black and Hyatt. (Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis 1969;99:696-702.) An electronic pressure transducer will be used (MicroRPM; Micromedical, Kent, UK) to register pressures. Reference values published by Rochester and Arora will be used to define percentages of normal respiratory muscle pressures. (Rochester DF, Arora NS. Respiratory muscle failure. Med Clin North Am 1983;67:573-97.)
Inspiratory Muscle Endurance during a constant load breathing task | Change from Baseline in endurance time at 8 weeks
  To measure inspiratory muscle endurance patients will be asked to breathe against a submaximal inspiratory load provided by a flow resistive loading device (POWERbreathe®KH1, HaB International Ltd., Southam, UK) until task failure. An inspiratory load will be selected that allows patients to continue breathing against the resistance for 3-7 minutes (typically between 50-60% of the Pi,max). Breathing instructions for patients will be the same as during the training sessions. Number of breaths, average duty cycle (inspiratory time as a fraction of the total respiratory cycle), average load, average power, and total work will be registered during the test by the handheld loading device. After 8 weeks of IMT the test will be repeated against an identical load and improvements in endurance time (seconds) will be registered as the main outcome. Changes in breathing parameters will be also registered.
Endurance capacity during a constant load cycling exercise test | Change from Baseline in endurance time at 8 weeks
  Endurance exercise testing will be conducted on an electronically braked cycle ergometer (Ergometrics 800S; SensorMedics, Anaheim, CA). This test will be performed at 75% of the peak work rate achieved during an incremental exercise test. Patients will be encouraged to continue exercising for as long as possible and upon exercise cessation they will be asked to verbalize their main reason for stopping exercise. Subjects will rate the magnitude of their perceived breathing and leg effort at rest, every 2 minutes during exercise and at end exercise by pointing to a 10-point Borg scale. Patients will also have to complete a questionnaire on descriptors of breathlessness at the end of the test. The test will be repeated against an identical intensity at the end of the training program. Changes in endurance time (sec) will be the main outcome.
Pulmonary Function | Change from Baseline in Pulmonary Function parameters at 8 weeks
  Pulmonary function Spirometry and whole body plethysmography will be performed according to the European Respiratory Society guidelines for pulmonary function testing (Vmax Autobox, Sensor Medics, Bilthoven, the Netherlands). (Quanjer PH, Tammeling GJ, Cotes JE, et al. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl 1993;16:5-40.) Changes in FEV1 (L), FVC (L), FRC (L), RV (L), IC (L) and peak inspiratory flow (L/s) will be registered.
Daily Physical Activity | Change in daily steps and time in moderate to vigorous daily physical activity from Baseline at 8 weeks
  Assessed with the SenseWear Pro3 activity monitor
Health related Quality of Life | Change from Baseline in health related quality of life at 8 weeks
  Assessed with the Saint George Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langer, Principal Investigator — KU Leuven
Locations (1):
- Queen's University, Kingston, Ontario, Canada